CLINICAL TRIAL: NCT01826110
Title: "[11C] PIB Comparison Study to [18F] AV-45 in Subjects With Alzheimer's Disease (AD) and Age Matched Healthy Controls"
Brief Title: PET Imaging Study Using [11C]PIB in Subjects With AD & Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NA_00033154; 1R21AG056142-01 (NIH)
Record Dates: First submitted 2013-02-22; First posted 2013-04-08 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [11C]PIB (Experimental): [11C]PIB
  Interventions: Drug: [11C]PIB

INTERVENTIONS:
Drug: [11C]PIB — Approximately 15 mCI [11C]PIB IV x1

SUMMARY:
The purpose of this study is to investigate the radiotracer [11C] PIB in participants with probably Alzheimer's Disease (AD) and healthy age-matched controls.

DETAILED DESCRIPTION:
The objectives of the study are:

1. To perform PET scans with [11C]PIB to use for direct (i.e., same-subjects) comparison of [11C]PIB and [18F]AV-45
2. To establish the most effective and reliable PET imaging method to detect amyloid deposition in AD, in order to understand disease progression and subsequently evaluate treatment effects.
3. To ascertain a PET imaging method that will minimize discomfort for subjects, thus increasing the potential for clinical follow-up scans, by reducing the patient burden and potential cost of future PET examinations.

A separate protocol/study will be conducted using [18F] AV-45. Participants who enroll in this protocol using [11C] PIB will be consented to participate in the [18F] AV-45 (IRB # NA_00033155) protocol/study as it is a mandatory requirement that participants participate in both protocols.Up to 20 participants with mild to moderate Alzheimer's Disease and 10 healthy volunteers will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years of age
* Subjects who in the opinion of the investigator based on medical history and physical exam can tolerate the PET scan procedures

Exclusion Criteria:

* Have clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances
* Have current clinically significant cardiovascular disease.
* Have a history of drug or alcohol abuse within the last year, or prior prolonged history of abuse
* Have a clinically significant infectious disease, including Acquired Immune Deficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV) infection or previous positive test for hepatitis
* Women of childbearing potential must not be pregnant (negative urine beta-hCG at the time of screening and negative urine beta-hCG on the day of imaging) or lactating at screening or at day of imaging
* Have a history of relevant severe drug allergy or hypersensitivity (Relevant severe drug allergies should be determined by the PI, and any questions about a subject's eligibility can be directed to Avid. If a subject has a history of severe drug allergies, it may be dangerous for them to participate in a study with a novel compound
* Have received an investigational medication within the last 30 days. Current clinically significant or unstable medical comorbidities, as indicated by history or physical exam
* Have received a radiopharmaceutical for imaging or therapy within the past 7 days prior to the imaging session for this study
* Body weight > 300 pounds
* History of significant radiation exposure
* Participants with pacemakers, implanted electronic hearing devices, aneurysm clips, shrapnel, unallowed prosthetic or other metallic device in their bodies
* Pre-existing CNS disease (other than dementia), endocrine, or severe cardiovascular disease (MI, CABG, angioplasty)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Distribution Volumes of 11C-PIB | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dean F Wong, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institution- Dept of Radiology , Division of Nuclear Medicine, Baltimore, Maryland, United States